CLINICAL TRIAL: NCT05219994
Title: Targeting the Carotid Bodies to Reduce Disease Risk Along the Diabetes Continuum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018486
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: After screening, participants will complete two study visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Glucose Tolerance Test (Experimental): Subjects will consume a 75 g glucose drink within 1-min and monitored for 2 hours.
  Interventions: Other: Hyperoxia Exposure; Other: Normoxia Exposure

INTERVENTIONS:
Other: Hyperoxia Exposure — 2 hours of hyperoxia exposure during OGTT
Other: Normoxia Exposure — 2 hours of normoxia exposure during OGTT

SUMMARY:
Our overall goal is to advance our understanding of the contribution of the carotid body chemoreceptors in glucose regulation and the development of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* healthy,
* type 2 diabetes
* BMI 18-40 kg/m2,
* non-pregnant,
* non-breastfeeding,
* non-nicotine users.

Exclusion Criteria:

* cardiovascular disease including myocardial infarction, heart failure, coronary artery disease, stroke;
* renal or hepatic diseases;
* active cancer;
* autoimmune diseases;
* immunosuppressant therapy;
* excessive alcohol consumption (>14 drinks/week);
* current nicotine use;
* foot ulcers;
* diabetic neuropathy;
* medication directly influencing sympathetic nervous system activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Glucose change in response to OGTT | 2 hours post glucose ingestion
Insulin change in response to OGTT | 2 hours post glucose ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Limberg, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided